CLINICAL TRIAL: NCT06055855
Title: A Randomized Controlled Trial Evaluating the Efficacy of Conventional Two-Needle Arthrocentesis Versus Surgery-Guided Arthrocentesis in the Management of Temporomandibular Joint Disorders
Brief Title: Comparing Two-Needle vs. Surgery-Guided Arthrocentesis for TMJ Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUDHF_FB_007
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Arthrocentesis,Temporomandibular Joint; Guided surgery
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Arthrocentesis Group (Active Comparator)
  Interventions: Procedure: Traditional Two-Needle Arthrocentesis
- Surgery-Guided Arthrocentesis Group (Experimental)
  Interventions: Procedure: Surgery-Guided Arthrocentesis

INTERVENTIONS:
Procedure: Traditional Two-Needle Arthrocentesis — Participants in this group will undergo arthrocentesis using the traditional two-needle technique. The procedure involves the placement of one or two needles into the temporomandibular joint (TMJ) to irrigate the joint space. Needle placement is guided by anatomical landmarks.
  Arms: Traditional Arthrocentesis Group
Procedure: Surgery-Guided Arthrocentesis — Participants in this group will receive arthrocentesis facilitated by a surgical guide. The guide is generated through pre-operative planning and is designed to aid in the accurate placement of the needle into the TMJ.
  Arms: Surgery-Guided Arthrocentesis Group

SUMMARY:
The goal of this clinical trial is to compare two methods of arthrocentesis in treating temporomandibular joint (TMJ) disorders. The main questions it aims to answer are:

Is surgery-guided arthrocentesis more efficient in terms of operation time compared to traditional two-needle arthrocentesis? Does the use of surgical guides lead to less postoperative pain and better patient comfort?

Participants will:

Undergo either the traditional two-needle arthrocentesis or the surgery-guided arthrocentesis.

Be monitored for operation time, postoperative pain, and overall patient comfort.

Researchers will compare the outcomes of patients who underwent traditional two-needle arthrocentesis with those who had surgery-guided arthrocentesis to see if the latter can shorten operation time and improve patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Wilkes stage II, III, or IV Temporomandibular Joint (TMJ) internal derangement.
* Presence of pain, sound, or both in the TMJ.
* Limitation or locking in mouth opening, or both.
* Patients who have not responded to symptoms after a minimum of three months of splint therapy.

Exclusion Criteria:

* Presence of infection in the puncture area.
* Presence of osteomyelitis in the neighboring region.
* Patients with uncontrolled coagulopathies.
* Patients experiencing limitation in maximum mouth opening without disk disorder.
* Patients with severe degenerative joint disease (e.g., deformed condylar contour, osteophyte findings in MRI).
* History of TMJ surgery.
* History of muscle-originated mandibular hypomobility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Total Duration of Arthrocentesis Procedure | Immediately following the completion of each arthrocentesis procedure, anticipated to occur on the day of the surgery.
  he primary outcome measure of the study is the total time duration required to complete the arthrocentesis procedure. This duration will be measured from the time local anesthesia is administered to the time when the arthrocentesis is completed. In addition, the number of intraoperative repositions of the needles will also be recorded.

SECONDARY OUTCOMES:
Volume of Ringer's Solution Used for Joint Irrigation | Immediately following the completion of each arthrocentesis procedure, anticipated to occur on the day of the surgery.
  The volume of Ringer's solution used to irrigate the temporomandibular joint during the arthrocentesis procedure will be measured.
Change in Postoperative Pain | 7 days
  Change in muscle pain intensity will be evaluated using a Visual Analogue Scale (VAS). The VAS comprises a 10 cm line, which can be presented either horizontally or vertically, anchored by "no pain" and "worst possible pain." Patients will be instructed to place a mark on the line that most accurately describes their level of muscle pain. These marks will be recorded and scored according to the VAS scale.
Change in Mouth Opening | 7 days
  The distance between the mesio-incisal corners of the upper and lower central incisors was measured with the help of a ruler when the mouth opening was at its maximum.
Change in Facial Swelling | 7 days
  With the technique described by Neupert ; Angle of mandible-tragus Angle of mandible-lateral canthus of eye Mandible corner-nose wing Angle of mandible oral-commissures Measurements were made with a tape measure from 5 points, with the mandible corner-pogonion.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided